CLINICAL TRIAL: NCT03114436
Title: Canada-DONATE: National Observational Study of Clinical Practices in Deceased Organ Donation
Brief Title: National Observational Study of Clinical Practices in Deceased Organ Donation
Acronym: CanadaDONATE
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Critical Care Trials Group (Other); Canadian National Transplant Research Program (Other); Transplant Quebec (Unknown); Trillium Gift of Life Network (Unknown); BC Transplant (Unknown); Southern Alberta Organ Donation Program (Unknown); Human Organ Procurement and Exchange (Unknown); Canadian Blood Services (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Maureen O. Meade, Research Program Director, McMaster University
Other Study IDs: Canada-DONATE 0780-PIA
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Deceased Organ Donation; Critical Illness; Transplantation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consented deceased organ donors: Includes neurological determination of death (DND) and by circulatory determination of death (DCD).
  Interventions: Other: Observational Data Collection

INTERVENTIONS:
Other: Observational Data Collection — All aspects of deceased donor care in the ICU.

SUMMARY:
This is a 1-year national prospective cohort study that observes the medical management of consented deceased organ donors at hospitals across Canada with a high volume of deceased donation.

DETAILED DESCRIPTION:
This prospective cohort study enrols consecutive adult deceased organ donors with a waiver of research consent and collects various data related to deceased donor care in the ICU from the time of consent for donation to the time of organ recovery. Clinical data includes donor characteristics, type of donation (after neurological death or cardiocirculatory death), resuscitation methods, cardiopulmonary monitoring techniques, medications, blood work, mechanical ventilation, diagnostic imaging, complications, and methods of death declaration. Various clinical data on deceased donors are collected prospectively from the time of consent for organ donation up to and including the day of organ recovery.

The Canada-DONATE study is designed to develop a national platform for future clinical trials in deceased donor care. The main objectives include:

1. Establish specialized organ donation research teams at participating ICUs.
2. Observe, record, and describe ICU practices in deceased donor care (e.g., donor resuscitation, organ suitability assessments, death declaration) which are likely to vary by site, region and province and will be very important to inform clinical care protocols for future RCTs.
3. Engage and work with ODOs from each province to foster data sharing and develop procedures to enhance efficiency in future RCTs.
4. Investigate the comparative effectiveness of various ICU interventions in deceased donor care to improve the conversion of consented donors to actual donors and to improve the number of transplants per donor.
5. Produce specific knowledge translation tools that will serve in the future as clinical tools to enhance ICU care and research tools to facilitate RCTs.

ELIGIBILITY:
Inclusion Criteria:

* Admitted into a critical care area (ICU, CCU, ER)
* Consent has been obtained for Organ Donation

Exclusion Criteria:

* Admitted into a paediatric critical care area (NICU, PICU)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients for whom consent for deceased organ donation has been obtained.
Sampling Method: Non-Probability Sample
Enrollment: 622 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence to national guidelines for deceased donor care | Duration of deceased donor care in the ICU (1-5 days per donor).
  For each donor, we will measure adherence to multiple recommendations from national guidelines for the management of deceased organ donors.

SECONDARY OUTCOMES:
Organ donation | Duration of deceased donor care in the ICU (1-5 days per donor).
  This refers to the conversion of a consented organ donor to an actual organ donor.
Organ transplantation | Transplantation may occur from 1-5 days from the time of consent.
  Deceased organ donors can provide up to 8 organ donations each. We will measure the number of transplants that proceed from each consented donor.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick D'Aragon, MD, MSc, Principal Investigator — Université de Sherbrooke; Maureen O Meade, MD, MSc, Study Director — McMaster University
Locations (29):
- Canada (29):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - Hamilton Health Sciences - Hamilton General Hospital, Hamilton, Ontario
  - Hamilton Health Science - Juravinski Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Trillium Health Partners - Trillium Health Centre, Mississauga, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital - General Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal - Hôpital Notre-Dame, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal - Hôtel-Dieu de Montréal, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal - Hôpital Saint-Luc, Montreal, Quebec
  - Centre Universitaire de Santé McGill/McGill University Health Centre - Hôpital Général de Montreal, Montreal, Quebec
  - Centre Universitaire de Santé McGill/McGill University Health Centre - Hôpital Royal Victoria, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Aragon F, Lamontagne F, Cook D, Dhanani S, Keenan S, Chasse M, English S, Burns KEA, Frenette AJ, Ball I, Boyd JG, Masse MH, Breau R, Akhtar A, Kramer A, Rochwerg B, Lauzier F, Kutsogiannis DJ, Ibrahim Q, Hand L, Zhou Q, Meade MO; Canadian Critical Care Trials Group and the Canadian Donation and Transplant Research Program. Variability in deceased donor care in Canada: a report of the Canada-DONATE cohort study. Can J Anaesth. 2020 Aug;67(8):992-1004. doi: 10.1007/s12630-020-01692-7. Epub 2020 May 8. PMID 32385825
- [Derived] D'Aragon F, Dhanani S, Lamontagne F, Cook DJ, Burns K, Akhtar A, Chasse M, Frenette AJ, Keenan S, Lize JF, Kutsogiannis DJ, Kramer A, Hand LE, Arseneau E, Masse MH, Ribic C, Ball I, Baker A, Boyd G, Rochwerg B, Healey A, Hanna S, Guyatt GH, Meade MO; Canadian Critical Care Trials Group and the Canadian National Transplant Research Program. Canada-DONATE study protocol: a prospective national observational study of the medical management of deceased organ donors. BMJ Open. 2017 Sep 28;7(9):e018858. doi: 10.1136/bmjopen-2017-018858. PMID 28963316
- See also: Canada-DONATE Research Progam Website — http://donate.ccctg.ca